CLINICAL TRIAL: NCT05926258
Title: A Prospective, Observer-blind, Randomized Clinical Trial to Investigate and Compare the Clinical Efficacy of Chloroprocaine 3% Gel and Oxybuprocaine 0.4% Eye Drops Anesthesia for Clinical Practice in Pediatric Population
Brief Title: Efficacy and Safety of Chloroprocaine 3% Gel and Oxybuprocaine 0.4% Eye Drops Anesthesia in Pediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHL.3-01-2021-M
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Local Anesthetic
Keywords: chloroprocaine; eye gel; ocular surface anesthesia
MeSH Terms: interventions — chloroprocaine; benoxinate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroprocaine 3% gel (Experimental): The assigned investigational product (2 drops) will be instilled in both eyes of each subject. Administrations will be performed at the clinical centre by the Investigator or his/her deputy on study day 1. For each administration, the 2 drops will be instilled one at the time, at a 1 min interval.
  Interventions: Drug: Chloroprocaine 3% eye gel
- Oxybuprocaine 0,4% solution (Active Comparator): The assigned active comparator (2 drops) will be instilled in both eyes of each subject. Administrations will be performed at the clinical centre by the Investigator or his/her deputy on study day 1. For each administration, the 2 drops will be instilled one at the time, at a 1 min interval.
  Interventions: Drug: Oxybuprocaine Hydrochloride 4 Mg/mL Eye Drops

INTERVENTIONS:
Drug: Chloroprocaine 3% eye gel — ocular surface anesthesia
  Other Names: Chemical Abstracts Service (CAS) nr 3858-89-7
  Arms: Chloroprocaine 3% gel
Drug: Oxybuprocaine Hydrochloride 4 Mg/mL Eye Drops — ocular surface anesthesia
  Other Names: Benoxinate
  Arms: Oxybuprocaine 0,4% solution

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of Chloroprocaine 3% eye gel compared to Oxybuprocaine 0,4% eye drops when used for inducing ocular surface anesthesia in pediatric patients.

74 Participants (male and female, aged 0-17 yrs) will be 1:1 randomized for receiving either the test drug (Chloroprocaine) or the reference drug (Oxybuprocaine) before undergoing to ocular exam who needs ocular surface anesthesia.

The successful surface anesthesia will be evaluated 5 minutes after receiving 2 drops (1 minute apart) of either test or reference drug by an eye spear sponge

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, patients must fulfil all these inclusion criteria:

1. Age ≥ one day of life (newborn, infant, child) and 17 years included (not anticipated to turn 18 during the study).
2. Female subjects currently either of:

   * Non-childbearing potential (i.e., premenarchal or physiologically incapable of becoming pregnant, including any female who is surgically sterilized via documented hysterectomy or bilateral tubal ligation), or
   * Childbearing potential (i.e., postmenarchal girls): the subject is eligible to enter and participate in this study if she is not lactating, has a negative pregnancy test and agrees to abstain from intercourses or uses a valid contraceptive method until study completion.
3. Signed written informed consent by both parents or legal representative(s) (unless only one has legal authority). Written informed assent for adolescents aged 12-17 years included and, whenever possible, informed assent for children aged 6 to 11 years included. Ability of the subjects and their parents/legal representative(s) to understand and comply with the protocol requirements, study-specified visit schedule and procedures.
4. Scheduled to undergo a routine clinical procedure which needs local ocular surface anesthesia, including but not limited to applanation tonometry, gonioscopy, Ultrasound Biomicroscopy (UBM), ocular ultrasonography, retinal peripheral examination with blepharostat and scleral indentation.

Exclusion Criteria:

* Patients fulfilling at the inclusion visit one or more of the following exclusion criteria will not be enrolled in the study:

Ophthalmic exclusion criteria

1. Previous ocular surgery less than 6 months before screening
2. Eye movement disorder (nystagmus)
3. History of herpetic keratitis
4. Corneal, epithelial, stromal or endothelial, residual or evolutionary disease (including corneal ulceration, corneal damage and superficial punctuate keratitis)
5. History of ocular traumatism, infection or inflammation within the last 3 months Systemic/non ophthalmic exclusion criteria

   • General history:
6. Any other medical or surgical history, disorder or disease such as acute or chronic severe organic disease: hepatic, endocrine neoplasia, hematological diseases, severe psychiatric illness, cardiac rhythm disorders and/or any complicating factor or structural abnormality judged by the investigator to be incompatible with the study

   • Allergic history:
7. Known hypersensitivity to one of the components of the investigational products Exclusion criteria related to general conditions
8. Non-compliant patient and/or parent(s)/legal representative(s) (e.g., not willing to attend the follow-up visits, way of life interfering with compliance)
9. Participation in another clinical study in the last three months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
10. Already included once in this study Exclusion criteria related to previous and concomitant medications / non-product therapies
11. Patient using any of the following previous and concomitant medication / treatment (according to the described periods) will not be included in the study:

NOT ALLOWED CONCOMITANT MEDICATIONS (washout times) Any change in concomitant anti-depressant medication: no changes permitted during the entire trial duration Any topical ocular treatment: within 15 days before inclusion Systemic opioids and morphine drugs, Sulohonamides, Anticholinesterase drugs: from 15 day before the inclusion visit onwards Any change in other systemic medication already ongoing before the inclusion visit: 7 days before the inclusion visit onwards Other systemic antalgics drugs (except for paracetamol)* from Day 1 onwards

*Paracetamol after primary endpoint assessment and oral, implantable, transdermal, or injectable contraceptives for child-bearing potential girls during the entire study will be allowed

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Conjunctiva anesthesia with Chloroprocaine 3% eye gel as compared with Oxybuprocaine chlorhydrate 0.4% eye drops | day 1
  Efficacy outcome: to assess the proportion of patients in each treatment group with a successful conjunctiva anesthesia in the right eye, 5 minutes after study product administration, i.e. right before the ocular examination, to be assessed by eye spear sponge.

SECONDARY OUTCOMES:
Assessing objective ocular signs | from day 1 until study end (day 8 or day 15)
  Evaluation of safety by assessing objective ocular signs (palpebral edema, chemosis, conjunctival hyperemia, conjunctival discharge, folliculo-papillary conjunctivitis, corneal staining punctations, anterior chamber cells, flare) and other objective ocular signs, assessed by slit lamp examination (SLE) or binocular indirect ophthalmoscopy (BIO), will be graded according to the following scale: 0=none, 1=mild, 2=moderate, 3=severe.
Occurrence of adverse events | from day 1 until study end (day 8 or day 15)
  Evaluation of safety by assessing the occurrence of adverse events throughout the study
Assessing the product global tolerance graded | day 1, post dose
  Evaluation of safety by assessing the product global tolerance graded by the Investigator by answering the following question "How do you consider the study product global tolerance" using the following scale: 0=very unsatisfactory, 1=unsatisfactory, 2= satisfactory, 3=very satisfactory.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Ospedale San Raffaele, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Ospedale della Donna e del Bambino, Ospedale Borgo Trento, Azienda Ospedaliera Universitaria Integrata, Verona, VR

IPD SHARING:
Plan to Share IPD: No